CLINICAL TRIAL: NCT03646487
Title: "Pro-Moms" - Mitigating the Effects of Structural Violence on Maternal Iron Status: a Randomized Placebo Controlled Pilot Study of Probiotic Supplementation in At-risk Pregnant Women
Brief Title: A Randomized Placebo Controlled Pilot Study of Probiotic Supplementation in At-risk Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary Dawn Koenig, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-0662; 5R34HL155481-03 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Iron-deficiency; Pregnancy, High Risk; Stress, Psychological
Keywords: pregnancy; iron status; structural violence
MeSH Terms: conditions — Anemia, Iron-Deficiency; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probiotic LP299v (Experimental): Women will receive 1 LP299v (10x10 colony forming units) in capsule form and 1 standard prenatal supplement in tablet form daily beginning at 15 weeks gestation through delivery.
  Interventions: Dietary Supplement: Probiotic LP299v 10x10 colony forming units in capsule form
- Placebo (Placebo Comparator): Women will receive 1 placebo in capsule form and 1 standard prenatal supplement in table form daily beginning at 15 weeks gestation through delivery.
  Interventions: Other: Placebo in capsule form

INTERVENTIONS:
Dietary Supplement: Probiotic LP299v 10x10 colony forming units in capsule form — Daily lactobacillus plantarum (LP299v) 10x10 colony forming units in capsule form
  Arms: Probiotic LP299v
Other: Placebo in capsule form — Daily placebo in capsule form
  Arms: Placebo

SUMMARY:
The goal of this randomized supplementation feasibility trial is to learn about the feasibility and preliminary efficacy of the probiotic, lactobacillus plantarum 299v (Lp299v), in pregnant individuals at-risk for iron deficiency anemia.

The main questions it aims to answer are:

* Is daily oral Lp299v a feasible and tolerable intervention for pregnant individuals to uptake?
* Does daily oral Lp299v in pregnancy impact maternal and neonatal cord hematological and iron status parameters?

Participants will be randomly assigned to one of two treatment groups: daily intake or probiotic Lp299v + prenatal vitamin with iron or placebo + prenatal vitamin with iron from 15-20 weeks of gestation through delivery.

Researchers will compare the two treatment groups to see if there is a difference in the feasibility of the intervention and the preliminary efficacy on maternal and neonatal cord hematological and iron status parameters.

DETAILED DESCRIPTION:
The most prevalent micronutrient deficiency in the United States (U.S.) is iron; a large majority of cases of iron deficiency (ID) and iron deficiency anemia (IDA) occur among pregnant women. During pregnancy, maternal iron stores are used for the growing fetus, maternal red blood cell (RBC) expansion, and placental growth and development, thus increasing the risk for ID and IDA. Across all trimesters of pregnancy in the U.S., it is estimated that 18% of individuals have ID and 5% have IDA, and within the third trimester, the prevalence of ID exceeds 27%. Prevalence of IDA is even greater among those who identify as Black or low-income. Maternal ID and IDA are associated with increased risk of preterm birth, low infant birth weight, maternal and fetal mortality, and irreversible infant neurocognitive defects. To meet this increasing requirement for iron and to optimize maternal iron nutrition, the Recommended Dietary Allowance for pregnancy is 27 mg/day of iron. However, given the continued high rates of maternal ID and IDA and only modest adherence to daily prenatal vitamins containing iron, alternative approaches to optimizing iron nutrition in pregnancy are needed.

Research has shown that one-time or short-term dosing of the probiotic Lactobacillus plantarum 299v (Lp299v) enhances iron absorption in non-pregnant populations. However, few studies have examined the effect of long-term supplementation on body iron stores. While probiotics are considered safe to consume in pregnancy, only one Lp299v supplementation trial has been conducted during the gestational period to evaluate its effects on maternal iron stores and risk of IDA. This study, among iron-sufficient pregnant Swedish women, showed a significantly lower decline in iron stores and a significantly lower prevalence of IDA in the third trimester among those randomized to Lp299v compared to standard care control.

These results offer potential positive effects for the role of Lp299v in maintaining maternal iron status among those starting pregnancy with sufficient iron stores and who receive care in a decentralized publicly funded healthcare system. However, no studies have evaluated the effect of Lp299v on maternal iron status among individuals at risk for IDA in pregnancy in the U.S., nor have studies extended findings to neonatal iron status. Moreover, it is unknown if positive feasibility and preliminary efficacy would persist in a U.S.-based health care setting with racially, ethnically, and socioeconomically diverse pregnant individuals. Therefore, the objectives of this study were as follows. First and foremost, we examined the feasibility of daily oral Lp299v maternal supplementation taken from the early second trimester through birth. Second, we explored the preliminary efficacy of Lp299v intake on maternal (at-risk for IDA defined as hemoglobin (Hb) between 10.0-12.0 g/dL) and neonatal cord hematological and iron status parameters compared to controls in an urban U.S. academic medical center with a racially, ethnically, and socioeconomically diverse patient population.

ELIGIBILITY:
Inclusion Criteria:

* a 1st trimester hemoglobin (Hb) of 10.0 - 11.9 g/dl demonstrating ID or risk for prenatal ID
* singleton
* naturally conceived pregnancy
* < 20 weeks gestation
* 18 - 45 years of age
* sufficient fluency in English to complete study forms
* refrain from non-study dietary and pre-/probiotic supplements while enrolled in the study

Exclusion Criteria:

* oral antibiotic use within the past 2 months
* autoimmune disease
* infection
* receiving steroid treatment
* bariatric surgery
* inflammatory bowel disease
* hyperemesis
* hematologic disorder (e.g., sickle cell disease)
* current tobacco use
* substance abuse in the last 6 months
* other chronic disorders such as type 2 diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dawn D Koenig, PhD, RN, CNM, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] OjiNjideka Hemphill N, Pezley L, Steffen A, Elam G, Kominiarek MA, Odoms-Young A, Kessee N, Hamm A, Tussing-Humphreys L, Koenig MD. Feasibility Study of Lactobacillus Plantarum 299v Probiotic Supplementation in an Urban Academic Facility among Diverse Pregnant Individuals. Nutrients. 2023 Feb 9;15(4):875. doi: 10.3390/nu15040875. PMID 36839232
- See also: Feasibility Study of Lactobacillus Plantarum 299v Probiotic Supplementation in an Urban Academic Facility among Diverse Pregnant Individuals — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9966742/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotic LP299v | Placebo
Started | 12 | 8
Completed | 7 | 6
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic LP299v | Placebo | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (6.5) | 28.7 (6.9) | 28.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 11 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20
Relationship status [Count of Participants; unit: Participants]
  Single not living with significant other | 5 | 2 | 7
  Single but living with significant other | 3 | 3 | 6
  Married | 4 | 3 | 7
Health insurance [Count of Participants; unit: Participants]
  Private | 6 | 1 | 7
  Public | 4 | 7 | 11
  Other | 2 | 0 | 2
Education [Count of Participants; unit: Participants]
  Some high school; some college | 9 | 7 | 16
  College graduate; graduate school | 3 | 1 | 4
Household income [Count of Participants; unit: Participants]
  ≤$30,999 | 7 | 7 | 14
  ≥$31,000 | 5 | 1 | 6
Receiving public assistance [Number; unit: participants]
  WIC (Women Infants and Children Program) | 3 | 2 | 5
  SNAP (Supplemental Nutrition Assistance Program) | 6 | 5 | 11
  TANF (Temporary Assistance for Needy Families) | 1 | 1 | 2
Gestational age at baseline [Mean (Standard Deviation); unit: weeks] | 12.6 (4.5) | 13.7 (3.7) | 13 (4.1)
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 38.6 (0.7) | 38.9 (0.7) | 38.8 (0.7)
Pre-pregnancy body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (7.3) | 31.8 (8.3) | 31.4 (7.5)
Pre-pregnancy obesity [Count of Participants; unit: Participants] | 7 | 4 | 11
Maternal body mass index (BMI) at baseline [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (6.8) | 32.9 (6.8) | 32.2 (6.7)
Maternal obesity at baseline [Count of Participants; unit: Participants] | 8 | 4 | 12
Parity [Count of Participants; unit: Participants]
  0 | 5 | 3 | 8
  1 | 3 | 3 | 6
  2 | 4 | 2 | 6
Food iron intake [Median (Inter-Quartile Range); unit: mg/1000 kcal] — Food iron intake was measured at baseline with a 24-hour diet recall (Nutrition Data System for Research (NDSR) software) using a multiple-pass interview approach, to standardize collection of the data.
  mg/1000 kcal | 11.2 [9.4 to 11.9] | 9.8 [8.3 to 25.4] | 10.5 [8.3 to 12.6]
Total iron (food and supplement) intake [Median (Inter-Quartile Range); unit: mg/1000 kcal] — Food iron intake was measured at baseline with a 24-hour diet recall (Nutrition Data System for Research (NDSR) software) using a multiple-pass interview approach, to standardize collection of the data. The consumption of dietary supplements was evaluated in concurrence with the 24-hour diet recall using the Dietary Supplement Assessment Module included in NDSR.
  mg/1000 kcal | 35.1 [18.1 to 39.8] | 36.8 [25.4 to 38.2] | 36.2 [18.5 to 38.6]

OUTCOME MEASURES:

1. Primary Outcome: Mean Adherence to the Supplement Regimen
Description: Mean adherence to the supplement regimen using Pillsy smart bottles and standard pill counts.
Time Frame: 15 weeks gestation through delivery, an average of 25 weeks
Population: A total of 20 participants were randomized in the study; n=12 in the Probiotic LP299v group and n=8 in the Placebo group. One participant in the Probiotic LP299v group completed the trial, but was not included in analysis because it was discovered the individual had alpha Thalassemia, a genetic disorder that impacts hemoglobin levels. Therefore, the overall number of participants analyzed in the Probiotic LP299v group was n=11.
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 11 | 8
percentage of adherence | 67 (29.1) | 80 (25.3)

2. Secondary Outcome: Number of Treatment-emergent Adverse Events Related to GI Symptoms
Description: Adverse events were captured using the Maternal Adherence Form beginning with the first pill refill visit through delivery. number of participants reporting adverse GI events
Time Frame: 15 weeks gestation through delivery, an average of 25 weeks
Population: as for outcome 1
Measure: Number; unit: GI events
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 11 | 8
GI events | 8 | 9

3. Secondary Outcome: Maternal Hemoglobin
Description: change in mean maternal serum hemoglobin (g/dl) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: We analyzed participants who completed the study with ≥80% adherence to examine changes in maternal hematological and iron status parameters by randomization group.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 4
g/dL | 0.4 [-1.1 to 1.8] | -0.1 [-1.7 to 1.6]

4. Secondary Outcome: Maternal Hematocrit
Description: Change in mean maternal serum hematocrit (%) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage by volume of red blood cells
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 4
percentage by volume of red blood cells | -0.03 [-6.6 to 6.5] | -0.5 [-4.7 to 3.8]

5. Secondary Outcome: Maternal Iron
Description: change in mean maternal serum iron (µg/dL) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: µg/dL
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
µg/dL | -5.2 [-17.6 to 7.2] | 5.7 [-48.8 to 60.2]

6. Secondary Outcome: Maternal Total Iron Binding Capacity
Description: change in mean maternal total iron binding capacity (µmol/L) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: µmol/L
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
µmol/L | 89.4 [12.4 to 166.4] | 58.3 [11.4 to 105.2]

7. Secondary Outcome: Maternal Serum Ferritin
Description: change in mean maternal serum ferritin (ng/mL) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
ng/mL | -4.4 [-9.4 to 0.6] | 0 [-94.4 to 94.4]

8. Secondary Outcome: Maternal Transferrin Saturation
Description: change in mean maternal transferrin saturation (%) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of saturation
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
percentage of saturation | -6.2 [-15.1 to 2.7] | -1.7 [-12.0 to 8.7]

9. Secondary Outcome: Maternal High-sensitivity C-reactive Protein (Hs-CRP)
Description: change in mean maternal high-sensitivity C-reactive protein (hs-CRP) (mg/L) from baseline to delivery
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
mg/L | -0.04 [-3.9 to 3.9] | -3.0 [-14.1 to 8.1]

10. Secondary Outcome: Maternal Iron Deficiency Anemia
Description: Number of participants who had iron deficiency anemia (IDA) at delivery. Hemoglobin, obtained from the Complete Blood Count, was used to define trimester-specific maternal IDA, with a downward correction of 0.8 g/dL for Black women. At the time of the study, it was recommended to use a race-adjusted cut-point for IDA. However, this race-adjusted cut-point was recently determined to be unfounded. IDA ranges included hemoglobin ≤11 g/dL for the first trimester, ≤10.5 g/dL for the second trimester, and ≤11 g/dL for the third trimester. IDA ranges with the correction for Black women were hemoglobin ≤10.2 g/dL for the first trimester, ≤9.7 g/dL for the second trimester, and ≤10.2 g/dL for the third trimester.
Time Frame: Assessed at baseline (i.e., 15-20 weeks gestation) through delivery; mean change from baseline to delivery is reported.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 1 | 2

11. Secondary Outcome: Infant Hemoglobin
Description: Mean infant serum hemoglobin (g/dl) from cord blood at delivery.
Time Frame: delivery
Population: The neonatal hematological and iron status parameters were examined for the newborns of mothers with ≥80% adherence to the supplement intervention.
Measure: Mean (95% Confidence Interval); unit: g/dl
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 4
g/dl | 14.7 [12.1 to 17.3] | 16.4 [14.6 to 18.2]

12. Secondary Outcome: Infant Hematocrit
Description: Mean infant serum hematocrit (%) from cord blood at delivery.
Time Frame: delivery
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: percentage by volume of red blood cells
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 4
percentage by volume of red blood cells | 44.3 [38.5 to 50.2] | 49.5 [44.9 to 54.0]

13. Secondary Outcome: Infant Iron
Description: Mean infant serum iron (µg/dL) from cord blood at delivery.
Time Frame: delivery
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: µg/dL
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
µg/dL | 136.2 [93.4 to 179.0] | 108.0 [48.4 to 167.6]

14. Secondary Outcome: Infant Total Iron Binding Capacity
Description: Mean infant total iron binding capacity (µmol/L) from cord blood at delivery.
Time Frame: delivery
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: µmol/L
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
µmol/L | 223.6 [155.6 to 291.6] | 274.0 [97.3 to 450.7]

15. Secondary Outcome: Infant Serum Ferritin
Description: Mean infant serum ferritin (ng/mL) from cord blood at delivery.
Time Frame: delivery
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
ng/mL | 88.8 [7 to 170.6] | 88.0 [44.1 to 132.0]

16. Secondary Outcome: Infant Transferrin Saturation
Description: Mean infant transferrin saturation (%) from cord blood at delivery.
Time Frame: delivery
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: percentage of saturation
Arm/Group | Probiotic LP299v | Placebo
Number analyzed (Participants) | 5 | 3
percentage of saturation | 63.8 [35.3 to 92.3] | 43.3 [-12.6 to 99.2]

ADVERSE EVENTS:
Time Frame: Health events were assessed by survey from the first pill refill visit through delivery, up to a period of 25 weeks span.
Description: Health events were assessed monthly by survey (i.e., Maternal Adherence Form) and through viewing provider notes in the participant's electronic health record. Study tolerability was defined a priori as no serious health events and the rate being similar between study arms. One participant in the Probiotic LP299v group completed the trial, but was not included in analysis due to alpha Thalassemia. Therefore, the overall number of participants analyzed in the Probiotic LP299v group was n=11.
Arm/Group | Probiotic LP299v | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 9/11 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic LP299v (N=11) | Placebo (N=8)
Genitourinary conditions (Reproductive system and breast disorders) | 4 (8) | 4 (5) — Genitourinary Conditions include vaginal yeast infection, short cervix, trichomonas, continuous urinary tract infection, chlamydia, frequent urination, vaginitis, and 'white stuff in urine'.
Gastrointestinal symptoms (Gastrointestinal disorders) | 8 (8) | 7 (9) — Gastrointestinal symptoms include abnormal oral glucose tolerance test, bloating, gassy, excessive stools, hemorrhoids, excessive saliva production, heart burn, nausea and food aversion.
Upper respiratory conditions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) — Upper Respiratory Conditions include shortness of breath, cold, asthma, sore throat.
Pain/swelling (General disorders) | 4 (8) | 5 (7) — Pain/Swelling includes back pain, round ligament pain, leg pain, carpal tunnel, and swelling.
Headaches/migraines (General disorders) | 3 (3) | 3 (3) — Categories include conditions as denoted by name.
Problems sleeping (General disorders) | 4 (4) | 4 (4) — Categories include conditions as denoted by name.
Emergency room visits (General disorders) | 2 (2) | 3 (3) — Categories include conditions as denoted by name.
Acne/rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Categories include conditions as denoted by name.
Anxiety/depression (Psychiatric disorders) | 2 (3) | 0 (0) — Categories include conditions as denoted by name.
Fatigue/tired (General disorders) | 5 (5) | 2 (2) — Categories include conditions as denoted by name.
Nosebleeds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) — Categories include conditions as denoted by name.
Genetic iron diagnoses (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) — Categories include conditions as denoted by name.
Genetic fetal diagnoses (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) — Categories include conditions as denoted by name.
Other (General disorders) | 1 (2) | 2 (2) — Other includes 'feeling warm', dizziness, and eyesight changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT03646487/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT03646487/ICF_001.pdf